CLINICAL TRIAL: NCT02539771
Title: Sleep Study in Adult Patients With Major Sickle Cell Disease With Paroxysmal Nocturnal Events
Acronym: DREPASOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P111121
Record Dates: First submitted 2015-07-27; First posted 2015-09-03 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Sickle Cell Disease
Keywords: vaso-occlusive crisis; obstructive sleep apnea; priapism
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Sleep Apnea, Obstructive; Priapism | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nocturnal VOC (Other)
  Interventions: Other: Polysomnography and blood sample
- Diurnal VOC (Other)
  Interventions: Other: Polysomnography and blood sample
- Slightly symptomatic (Other)
  Interventions: Other: Polysomnography and blood sample

INTERVENTIONS:
Other: Polysomnography and blood sample — Blood collection is a specific intervention of protocol for the 3 arms. Polysomnography is a specific intervention for the arms " Diurnal VOC " and " Slightly symptomatic "

SUMMARY:
Hypothesis is that the occurrence of nocturnal Vaso-Occlusive Crisis (VOC) and priapism in adults might be related to episodes of nocturnal desaturation secondary to a sleep apnea syndrome. Investigator hypothesize that chronic biological consequences of Obstructive Sleep Apnea (hypercoagulability, endothelial dysfunction ...) favour VOC and acute manifestations (nocturnal desaturation) favour nocturnal VOC.

The confirmation of this hypothesis will lead investigator to propose a systematic screening of obstructive sleep apnea (OSA) in patients with nocturnal VOC. Moreover, systematic treatment of OSA in sickle cell patients could help significantly reduce the number and severity of nocturnal VOC.

ELIGIBILITY:
Inclusion Criteria:

Night VOC Group:

* night VOC ≥ 2 in the previous year
* written informed consent

Daytime VOC Group:

* VOC no nocturnal
* diurnal VOC ≥ 2 in the previous year
* written informed consent

Slightly symptomatic group:

* no hospitalization for VOC
* written informed consent

Exclusion Criteria:

* Taking opioids
* Taking medication that alters sleep (antidepressants, benzodiazepines ...)
* Known history of sleep apnea syndrome
* Known history of serious psychiatric disorder
* Recent vaso-occlusive crisis (within 3 weeks)
* Changes in background treatment (Hydrea or exchange transfusions) in the past 12 months
* Inactive affiliation to social security
* Under legal protection
* A female who is pregnant or breastfeeding
* Prisoners
* Emergency situation
* Refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with nocturnal desaturation and patients with OSA | at 1 year

SECONDARY OUTCOMES:
Oxygen desaturation index | at 1 year
Minimum oxygen saturation level | at 1 year
Quantitative analysis of biomarkers in plasma samples | at 1 year
Quantitative analysis of proinflammatory and anti-inflammatory cytokines | at 1 year
Minimum oxygen saturation level during rapid eye movement (REM) sleep in patients with recurrent priapism and in patients who never presented priapism | at 1 year
Apnea-Hypopnea Index | at 1 year
Sleep time with arterial oxygen saturation less than 90% | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anoosha Habibi, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWNED BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION